CLINICAL TRIAL: NCT00262834
Title: A Pilot Study Evaluating Surrogates of Response to Short Term Oral Suberoylanilide Hydroxamic Acid (SAHA) in Women With Newly Diagnosed Breast Cancer
Brief Title: Vorinostat in Treating Women Who Are Undergoing Surgery For Newly Diagnosed Stage I -III Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00098; NCI-2009-00098 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000445404 (Other: Clinical Data Repository (CT.gov)); SKCCC J0504 (Other: Johns Hopkins University/Sidney Kimmel Cancer Center); 6914 (Other: CTEP); U01CA070095 (NIH); P30CA006973 (NIH)
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer; Stage I Breast Cancer; Stage II Breast Cancer; Stage III Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Vorinostat; Surgical Procedures, Operative; Congresses as Topic

STUDY DESIGN:
Intervention Model Description: Patients receive oral vorinostat twice daily on days -3 to 0. Approximately 2 hours after the final dose of vorinostat, patients undergo conventional surgical resection of the tumor on day 0. After completion of study treatment, patients are followed for 30 days.

ARMS (1):
- Arm I (Experimental): Patients receive oral vorinostat twice daily on days -3 to 0. Approximately 2 hours after the final dose of vorinostat, patients undergo conventional surgery of the tumor on day 0. After completion of study treatment, patients are followed for 30 days.
  Interventions: Drug: vorinostat; Other: conventional surgery

INTERVENTIONS:
Drug: vorinostat — Given orally, conventional surgery to follow.
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Other: conventional surgery — Undergo conventional surgery
  Other Names: surgery, conventional

SUMMARY:
This phase II trial is studying how well vorinostat works in treating women who are undergoing surgery for newly diagnosed stage I, stage II, or stage III breast cancer. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving vorinostat before surgery may shrink the tumor so that it can be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the safety and tolerability of vorinostat in women undergoing conventional surgery for newly diagnosed stage I-III breast cancer.

OULINE: This is a multicenter, pilot study.

Patients receive oral vorinostat twice daily on days -3 to 0. Approximately 2 hours after the final dose of vorinostat, patients undergo surgical resection of the tumor on day 0.

After completion of study treatment, patients are followed for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* No prior or concurrent hormonal therapy for breast cancer
* Histologically confirmed breast cancer, stage I-III disease, scheduled to undergo definitive surgery or other primary treatment (e.g., preoperative/neoadjuvant systemic treatment) for breast cancer
* ECOG 0-2 OR Karnofsky 60-100%
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal
* PT ≤ 14 seconds
* Creatinine normal
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled intercurrent illness
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to vorinostat
* At least 30 days since prior hormone replacement therapy (e.g., estrogen and/or progestin)
* Concurrent vaginal hormone preparations (e.g., vagifem or estring) allowed
* No concurrent birth control pills
* No prior radiotherapy to the ipsilateral breast
* No prior or concurrent radiotherapy for breast cancer
* No prior or concurrent novel therapy for breast cancer
* At least 14 days since prior valproic acid or another histone deacetylase inhibitor
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent therapy for this cancer
* WBC ≥ 3,000/mm^3

Exclusion criteria:

* Patients must not be recieving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to SAHA.
* Patients may not be taking valproic acid or another histone deacetylase inhibitor for at least 2 weeks prior to initiating SAHA.
* Women who are pregnant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2005-10; Primary Completion 2008-10 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vered Stearns, Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (1):
- Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women enrolled from two sites, Johns Hopkins Medical Institutes and Anne Arundel Medical Center. Informed consent was obtained from all participants in the vorinostat and control groups.
Pre-assignment Details: Women must have adequate performance status and blood counts/organ function; no hormones within 30 days of diagnostic biopsy, prior or concomitant treatment for the current cancer, or uncontrolled intercurrent illness that could limit compliance were allowed.
Groups:
- Vorinostat: Women in the vorinostat group were scheduled to receive 6 doses of oral vorinostat at 300 mg twice daily (bid), with the last dose administered by study personnel approximately 2 hours before the scheduled breast surgery (or biopsy).
- Tissue Only: Women who declined vorinostat but agreed to donate tissues for biomarker assessment, signed a separate informed consent and were enrolled as controls.
Period: Overall Study
Arm/Group | Vorinostat | Tissue Only
Started | 25 | 29
Completed | 24 | 25
Not Completed | 1 | 4
Not completed — Surgery delayed/tissue not collected | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vorinostat | Tissue Only | Total
Number analyzed (Participants) | 25 | 29 | 54
Age, Continuous [Median (Full Range); unit: years] | 55 [34 to 71] | 52 [34 to 79] | 54 [34 to 79]
Age, Customized [Number; unit: years]
  <=18 years | 0 | 0 | 0
  >18 years | 25 | 29 | 54
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 29 | 54
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 29 | 54

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Participants were evaluated for adverse events due to vorinostat to assess if it was safe to give the drug prior to surgery. 17 of 25 participants who received vorinostat experienced at least 1 adverse event believed to be related to the study drug; no adverse events were severe, and the treatment was considered safe.
Time Frame: After 3 days of vorinostat
Population: Participants who received at least one dose of vorinostat.
Measure: Number; unit: participants
Arm/Group | Vorinostat
Number analyzed (Participants) | 25
participants | 17

2. Primary Outcome: Change in Tissue Proliferation After 3 Days of Treatment
Description: Change in Ki-67 (a marker of tissue proliferation) by IHC compared to baseline in the treated (22 evaluable samples) or untreated patients (15 evaluable samples) were analyzed between groups. Ki-67 is a protein in cells that increases as cellsprepare to divide into new cells. A staining process can measure the percentage of tumor cells that are positive for Ki-67. The more positive cells there are, the more quickly they are dividing and forming new cells.
Time Frame: After 3 days of vorinostat
Population: Matched samples (ie, diagnostic biopsy and surgical tissues) for Ki-67 by IHC were available from 22 (92%) treated and from 15 (60%) controls.
Measure: Mean (Full Range); unit: percentage of change
Units Other Than Participants: Evaluable tissue samples
Arm/Group | Vorinostat | Tissue Only
Number analyzed (Participants) | 25 | 29
Number analyzed (Evaluable tissue samples) | 22 | 15
percentage of change | -3 [-62 to 38] | -4 [-32 to 46]
Statistical Analysis 1: Comparison: Vorinostat vs Tissue Only; Test type: Superiority or Other; p = 0.42, Wilcoxon (Mann-Whitney); Wilcoxon rank-sum tests were used to compare the differences (post-pre) between groups

3. Primary Outcome: Change in Tissue Apoptosis After 3 Days of Treatment
Description: Change in cleaved caspase-3 (a marker of tissue apoptosis) by IHC compared to baseline in the treated (19 evaluable samples) or untreated patients (12 evaluable samples) were analyzed between groups. Cleaved caspase-3 is a protein in cells involved in apoptosis (cell death).
Time Frame: Baseline and after 3 day of vorinostat
Population: Matched samples (ie, diagnostic biopsy and surgical tissues) for cleaved caspase-3 by IHC were available from 19 (71%) treated and from 12 (48%) controls.
Measure: Mean (Full Range); unit: percentage of change
Units Other Than Participants: Evaluable tissue samples
Arm/Group | Vorinostat | Tissue Only
Number analyzed (Participants) | 25 | 29
Number analyzed (Evaluable tissue samples) | 19 | 12
percentage of change | 0 [-5 to 5] | 0 [-2 to 3]
Statistical Analysis 1: Comparison: Vorinostat vs Tissue Only; Test type: Superiority or Other; p = 0.50, Wilcoxon (Mann-Whitney); Wilcoxon rank-sum tests were used to compare the differences (post-pre) between groups

4. Secondary Outcome: Change in Tissue Histone Acetylation After 3 Days of Treatment
Description: To evaluate change from baseline in tissue histone acetylation in patients with primary breast cancer who received three days of Short Term Oral Suberoylanilide Hydroxamic Acid (SAHA) 300 mg PO bid immediately prior to definitive breast surgery or other primary treatment. This is measured by Cumulative Methylation Index, which is reported as the sum of all %M for all genes. %M= (methylated copies divided by methylated + unmethylated copies) x 100.
Time Frame: Baseline and after 3 day of Vorinostat
Population: 25 matched samples were collected; however, only 19 were available for analysis as there were 6 cases that were not evaluable for Cumulative Methylation Index.
Measure: Number; unit: Cumulative Methylation Index
Arm/Group | Arm I
Number analyzed (Participants) | 19
Cumulative Methylation Index | 38.3
Statistical Analysis 1: Comparison: Arm I; Test type: Other; p = 0.24, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Blood (Peripheral Blood Mononuclear Cells) Histone Acetylation After 3 Days of Treatment
Description: To evaluate baseline and change in histone acetylation in polymononuclear cells in patients with primary breast cancer who received three days of SAHA 300 mg PO bid immediately prior to definitive breast surgery or other primary treatment.
Time Frame: Baseline and after 3 day of Vorinostat
Population: No data was collected for this outcome. We were not able to successfully dissolve the pellet in lysis buffer, and the samples were not subjected to histone acetylation analyses.
Arm/Group | Vorinostat | Tissue Only
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline and after 3 day of vorinostat
Description: Participants were assessed by study staff a specified time points per CTCAE 3.0.
Groups:
- Vorinostat: Women in the vorinostat group were scheduled to receive 6 doses of oral vorinostat at 300 mg twice daily (bid), with the last dose administered by study personnel approximately 2 hours before the scheduled breast surgery (or biopsy).
  Only vortinostat group adverse events were reported or collected to assess association of events with the agent in question.
Arm/Group | Vorinostat
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 17/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat (N=25)
Diarrhea (Gastrointestinal disorders) | 7 (7)
Fatigue (General disorders) | 4 (4)
Dysgeusia (Gastrointestinal disorders) | 4 (4)
Anorexia (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (4)
Headache (Nervous system disorders) | 1 (1)
White blood cell decreased (Investigations) | 6 (6)

LIMITATIONS AND CAVEATS:
The main limitation of the trial is the unexpectedly low proportion of matched evaluable samples available for the biomarkers studied, ranging from 44% to 92%.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less